CLINICAL TRIAL: NCT00454961
Title: Effectiveness of Artemether-Lumefantrine Treatment Provided by Community Health Worker Against Uncomplicated Malaria in Children Under 5 Years of Age in Tanzania
Brief Title: Effectiveness of Artemether-Lumefantrine for Malaria Treatment of Children at Community Level in Tanzania
Acronym: C3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCC-2007
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; artemether-lumefantrine; effectiveness
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: artemether-lumefantrine

SUMMARY:
The purpose of this clinical trial is to assess the effectiveness of artemether-lumefantrine (Coartem®) treatment provided by community health workers against uncomplicated malaria in children under 5 years of age in Kibaha District, Tanzania, during an extended follow-up of 42 days. The hypothesis is that artemether-lumefantrine treatment provided by community health workers will result in less than 85% PCR-corrected parasitological effectiveness by day 42, mainly due to partial non-compliance to full standard 6-dose regimen of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Aged <5 years
2. Weight >5 kg
3. Suffering from acute uncomplicated P. falciparum malaria confirmed by RDT. Later microscopy using Giemsa-stained thick film will be made to ensure asexual parasite density of 2000 to 200 000 parasites/µL
4. Having a history of fever in the preceding 24 h
5. Able to ingest tablets orally
6. Willing and able to attend stipulated follow-up visits
7. With written informed consent from parent/guardian for children to participate in the trial.

Exclusion Criteria:

Presenting with any of the following "danger signs of severe malaria":

1. Convulsions (>1 episode within previous 24 hours)
2. Lethargic/unconscious

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2007-04

PRIMARY OUTCOMES:
Effectiveness (PCR adjusted parasitological cure rate) of artemether-lumefantrine
during 42 days follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, Professor, Study Director — Karolinska University Hospital
Locations (1):
- Kibaha District, Kibaha, Tanzania

REFERENCES:
- [Derived] Ngasala BE, Malmberg M, Carlsson AM, Ferreira PE, Petzold MG, Blessborn D, Bergqvist Y, Gil JP, Premji Z, Martensson A. Effectiveness of artemether-lumefantrine provided by community health workers in under-five children with uncomplicated malaria in rural Tanzania: an open label prospective study. Malar J. 2011 Mar 16;10:64. doi: 10.1186/1475-2875-10-64. PMID 21410954